CLINICAL TRIAL: NCT00923559
Title: A Randomized Controlled Trial of Mother-Infant Psychoanalytic Treatment (MIP) and Treatment As Usual (TAU) at Child Health Centres (CHC)
Brief Title: Mother-Infant Psychoanalysis Project of Stockholm
Acronym: MIPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Bjorn Salomonsson, Doct. student, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIPPS-01
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Mother-infant Relational Disturbances
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mother-Infant Psychoanalytic treatment;MIP (Experimental): MIP intervention
  Interventions: Other: Mother-Infant Psychoanalytic treatment (MIP)
- TAU at Child Health Centres (Active Comparator): Regular nurse visits at Child Health Centres according to Swedish infant health care.
  Interventions: Other: Treatment as Usual at Child Health Centre

INTERVENTIONS:
Other: Treatment as Usual at Child Health Centre — Treatment as usual (TAU) involved scheduled nurse calls at the local Child Health Centre (CHC), with paediatric checkups at 2 and 6 months of age. The nurse is encouraged to promote attachment and to detect postnatal depressions. Mothers might be offered parental groups, infant massage or guidance promoting interaction, as well as appointments with a paediatrician or a child psychiatric psychologist. Within the TAU framework, additional treatment might be initiated by the nurse or the mother. This was registered at the end-point interview.
  Arms: TAU at Child Health Centres
Other: Mother-Infant Psychoanalytic treatment (MIP) — MIP (Norman, 2001; 2004) is a psychoanalytic method adapted to the requirements of the infant as analysand in the presence of his mother. In the study, the analysts strived to recruit the baby for an emotional interchange, though this did not imply any belief that the infant would understand verbal communication. Rather, the analyst addressed the baby to help him liberate emotions consolidated in symptoms such as screaming, avoiding maternal eye contact, and breast refusal. The analyst took care in enrolling the participant mother. This was to enhance her understanding of the baby's predicament and the nature of their relation, as well as giving her space to vent her own frustration, depression and anxiety.
  Arms: Mother-Infant Psychoanalytic treatment;MIP

SUMMARY:
Mother-infant relationship disturbances broadly comprise three areas; maternal distress, infant functional problems, and relationship difficulties. Given the high frequency of such disturbances and the relative paucity of randomized treatment studies, substantial systematic investigation is needed. This project is a randomized controlled study comparing mother-infant psychoanalytic treatment with treatment as usual in cases where mothers and/or health visitors demanded expert help.

DETAILED DESCRIPTION:
DESIGN

Eighty dyads with infants below 1½ years of age were interviewed and then randomly assigned to MIP or TAU. An end-point interview followed after ½ year, evaluating the intervention effects.

The MIP treatments were performed by IPA psychoanalysts at the Infant Reception Service of the Swedish Psychoanalytic Society. TAU implied contact with a nurse at a Child Health Centre, as part of regular Swedish health care of infants and mothers. Additional treatments within the TAU framework suggested at the initiative by the health visitor or the mother were registered at the end-point interview.

INSTRUMENTS

Mother-report questionnaires; the Ages and Stages Questionnaire:Social-Emotional (ASQ:SE; Squires et al., 2002), the Edinburgh Postnatal Depression Scale (EPDS; Cox et al., 1987), the General Severity Index of the Symptom Check List-90 (Derogatis, 1994)and the Swedish Parental Questionnaire (SPSQ; Östberg et al., 1997).

Time frame: All four instruments were measured at intake interviews and six months later.

Independently rated video-taped mother-infant interactions: the Emotional Availability Scale (EAS; Biringen, 1998).

Relationship assessment: the Parent-Infant Relationship Global Assessment Scale (PIR-GAS; ZERO-TO-THREE, 2005).

ELIGIBILITY:
Inclusion Criteria:

* The mother expressed significant concerns about one or more of the following domains: herself as a mother, her infant's well-being, or the mother-baby relationship (this was operationalized as a score < 80 ("perturbed relation") on the PIR-GAS or, alternatively, > 2.5 on the SPSQ).
* Infant of any gender, age below 18 months.
* Duration of worries exceeding two weeks.
* Domicile in Stockholm.
* Reasonable mastery of Swedish.

Exclusion Criteria:

* Maternal psychosis.
* Substance dependence according to DSM-IV, to an extent precluding collaboration.

No mothers met these criteria.

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per-Anders Rydelius, Professor, Study Director — Karolinska Institutet
Locations (1):
- Karolinska Institute, Stockholm, Sweden

REFERENCES:
- [Background] Salomonsson B. "Talk to me baby, tell me what's the matter now". Semiotic and developmental perspectives on communication in psychoanalytic infant treatment. Int J Psychoanal. 2007 Feb;88(Pt 1):127-46. doi: 10.1516/04p3-fuer-0u41-lln8. PMID 17244571
- [Background] Salomonsson B. Semiotic transformations in psychoanalysis with infants and adults. Int J Psychoanal. 2007 Oct;88(Pt 5):1201-21. doi: 10.1516/ijpa.2007.1201. PMID 17908677
- [Background] Salomonsson B, Sleed M. The Ages & Stages Questionnaire: Social-Emotional: A validation study of a mother-report questionnaire on a clinical mother-infant sample. Infant Ment Health J. 2010 Jul;31(4):412-431. doi: 10.1002/imhj.20263. PMID 28543080
- [Background] Salomonsson, B. (2009). Mother-infant work and its impact on psychoanalysis with adults. Scandinavian Psychoanalytic Review, 32, 3-13.
- [Background] Salomonsson B. The music of containment: Addressing the participants in mother-infant psychoanalytic treatment. Infant Ment Health J. 2011 Nov;32(6):599-612. doi: 10.1002/imhj.20319. Epub 2011 Nov 3. PMID 28520149
- [Result] Salomonsson B, Sandell R. A randomized controlled trial of mother-infant psychoanalytic treatment: I. Outcomes on self-report questionnaires and external ratings. Infant Ment Health J. 2011 Mar;32(2):207-231. doi: 10.1002/imhj.20291. PMID 26908296
- [Result] Salomonsson B, Sandell R. A randomized controlled trial of mother-infant psychoanalytic treatment: II. Predictive and moderating influences of qualitative patient factors. Infant Ment Health J. 2011 May;32(3):377-404. doi: 10.1002/imhj.20302. PMID 26904966
- See also: Describes the research project and its clinical utility in lay language — http://www.bjornsalomonsson.se

RESULTS

PARTICIPANT FLOW:
Groups:
- Mother-Infant Psychoanalytic Treatment;MIP: MIP (Norman, 2001; 2004) is a psychoanalytic method adapted to the requirements of the infant as analysand in the presence of his mother. The analyst strives to recruit the baby for an emotional interchange, though this does not imply any belief that the infant understands verbal communication. The analyst addresses the baby to help him liberate emotions consolidated in symptoms such as screaming, avoiding maternal eye contact, and breast refusal. The analyst also enrolls the participant mother. This is to enhance her understanding of the baby's predicament and the nature of their relation, as well as giving her space vent her frustration, depression and anxiety.
- TAU at Child Health Centres: Scheduled nurse calls at the local Child Health Centre (CHC), with paediatric checkups at 2 and 6 months of age. The nurse is encouraged to promote attachment and to detect postnatal depressions. Mothers may be offered parental groups, infant massage or guidance promoting interaction, as well as appointments with a paediatrician or a child psychiatric psychologist. Within the CHC framework, additional treatment may initiated by the nurse or the mother. This will be registered at the end-point interview.
Period: Overall Study
Arm/Group | Mother-Infant Psychoanalytic Treatment;MIP | TAU at Child Health Centres
Started | 40 | 40
Completed | 38 | 37
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mother-Infant Psychoanalytic Treatment;MIP | TAU at Child Health Centres | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (3.5) | 32.3 (4.6) | 33.2 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: The Parent-Infant Relationship Global Assessment Scale (PIR-GAS; ZERO-TO-THREE, 2005)
Description: An observer-rated scale ranging from 0 to 99, from "documented maltreatment" to "well-adapted". Higher scores indicate a better outcome. Inter-rater reliability was measured with an external experienced infant psychotherapist.
Time Frame: Two interviews, six months apart
Population: Outliers (z-transformed scores>3.29) were replaced by raw scores corresponding to z=3.29. Multivariate outliers identified via Mahalanobi's distance through a multiple regression, none found. Missing data were very rare and missing at random. No scores imputed. Intention to treat (ITT)analysis was used.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- Mother-Infant Psychoanalytic Treatment;MIP: A psychoanalytic method adapted to the requirements of the infant as analysand in the presence of his mother. The analyst recruits the baby for an emotional interchange, though this does not imply any belief that the infant understands verbal communication. The analyst addresses the baby to help him liberate emotions consolidated in symptoms such as screaming, avoiding maternal eye contact, and breast refusal. The analyst also enrolls the participant mother to enhance her understanding of the baby's predicament and the nature of their relation, as well as giving her space to vent her own frustration, depression and anxiety.
- Treatment as Usual at Child Health Centre: Treatment as usual with nurse visits at Child Health Centres as part of regular Swedish child health care.
Arm/Group | Mother-Infant Psychoanalytic Treatment;MIP | Treatment as Usual at Child Health Centre
Number analyzed (Participants) | 38 | 37
Scores on a scale | 83.53 [79.56 to 87.50] | 76.67 [72.74 to 80.60]
Statistical Analysis 1: Comparison: Mother-Infant Psychoanalytic Treatment;MIP vs Treatment as Usual at Child Health Centre; Null hypothesis: MIP and CHC care should yield equal outcomes. For power calculations, studies on the EPDS and the SPSQ were used. An estimated power of .80 and a two-tailed significance of .05 would necessitate between 29 and 60 participants. Forty dyads per group were chosen; Test type: Superiority or Other; p = .006, Regression, Linear — Null hypothesis MIP and CHC care should yield equal outcomes. A priori threshold p<.05; Degrees of freedom (df) = 68.3; Mean Difference (Final Values) = 8.69, 95% CI [2.64 to 14.74], Standard Error of Mean 3.04

2. Primary Outcome: the Edinburgh Postnatal Depression Scale (EPDS; Cox et al., 1987)
Description: The EPDS (Swedish translation, Lundh & Gylland, 1990), is a self-report questionnaire containing 10 items each with a 3-point scale. Range: 0 - 30. Higher scores indicate a worse outcome. It is widely used at Swedish CHCs and has been validated on samples in Sweden.
Time Frame: Two interviews, six months apart
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- Treatment as Usual at Child Health Centres: Treatment as usual with nurse visits at Child HEalth Centres as part of regular Swedish child health care.
Arm/Group | Mother-Infant Psychoanalytic Treatment;MIP | Treatment as Usual at Child Health Centres
Number analyzed (Participants) | 38 | 37
Scores on a scale | 6.28 [4.82 to 7.74] | 7.99 [6.56 to 9.43]
Statistical Analysis 1: Comparison: Mother-Infant Psychoanalytic Treatment;MIP vs Treatment as Usual at Child Health Centres; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .018, Regression, Linear — p-value unadjusted for multiple comparisons. A priori threshold p<.05; Degrees of freedom (df) = 69.3; Mean Difference (Final Values) = 2.57, 95% CI 2-sided [0.46 to 4.68], Standard Error of Mean 1.06

3. Primary Outcome: the Ages and Stages Questionnaire: Social-Emotional, (ASQ:SE; Squires et al., 2002
Description: Items are mostly rated on a 4-step scale, with 0,5,10 or 15 points per item, where 0 is most optimal. There are three versions for the age ranges of this study: 3-8, 9-14, and 15-20 months. To enable comparison across age groups we report mean scores across all items. Higher scores indicate a worse outcome. Each version was independently translated into Swedish, retranslated and approved by the constructor.
Time Frame: Two interviews, six months apart
Population: Outliers (z-transformed scores>3.29) were replaced by raw scores corresponding to z=3.29.Multivariate outliers identified via Mahalanobi's distance through a multiple regression, none found. Missing data were very rare and missing at random. No scores imputed. Intention to treat (ITT)analysis was used.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- Mother-infant Psychoanalytic Treatment; MIP: A psychoanalytic method adapted to the requirements of the infant as analysand in the presence of his mother. The analyst recruits the baby for an emotional interchange, though this does not imply any belief that the infant understands verbal communication. The analyst addresses the baby to help him liberate emotions consolidated in symptoms such as screaming, avoiding maternal eye contact, and breast refusal. The analyst also enrolls the participant mother to enhance her understanding of the baby's predicament and the nature of their relation, as well as giving her space to vent her own frustration, depression and anxiety.
Arm/Group | Mother-infant Psychoanalytic Treatment; MIP | Treatment as Usual at Child Health Centres
Number analyzed (Participants) | 38 | 37
Scores on a scale | 1.00 [0.77 to 1.24] | 1.14 [0.90 to 1.37]
Statistical Analysis 1: Comparison: Mother-infant Psychoanalytic Treatment; MIP vs Treatment as Usual at Child Health Centres; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .266, Regression, Linear — p-value unadjusted for multiple comparisons. A priori threshold p<.05; Degrees of freedom = 73.4; Mean Difference (Net) = 0.27, 95% CI 2-sided [-0.21 to 0.75], Standard Error of Mean 0.24

4. Secondary Outcome: the Swedish Parental Stress Questionnaire, (SPSQ; Östberg et al., 1997)
Description: A Swedish-language version of the Parenting Stress Index (PSI; Abidin, 1990) with 35 items, each ranging 1-5 points. Higher scores indicate a worse outcome.
Time Frame: Two interviews six months apart
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Mother-Infant Psychoanalytic Treatment;MIP | Treatment as Usual at Child Health Centres
Number analyzed (Participants) | 38 | 37
Scores on a scale | 2.67 [2.50 to 2.85] | 2.74 [2.57 to 2.91]
Statistical Analysis 1: Comparison: Mother-Infant Psychoanalytic Treatment;MIP vs Treatment as Usual at Child Health Centres; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .052, Regression, Linear — p-value unadjusted for multiple comparisons. A priori threshold p<.05; Mean Difference (Net) = 0.16, 95% CI 2-sided [0.00 to 0.32], Standard Error of Mean 0.08

5. Secondary Outcome: the Emotional Availability Scales, Subscale on Sensitivity (EAS; Biringen, 1998)
Description: The EAS assessed video-taped mother-baby interactions of 10' duration on three maternal dimensions (Sensitivity, Structuring, Non-intrusiveness) and two infant dimensions (Responsiveness and Involvement. The raw scores of the subscales have different ranges (0-5, 0-7, and 0-9). To enable comparison across subscales, we divided scores in each subscale with its maximal score. This yielded a range for each subscale of 0-1.Thus, the total score range for all subscales was 0-1, with higher scores indicating a better outcome. Here we report results on Sensitivity.
Time Frame: Two interviews, six months apart
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mother-infant Psychoanalytic Treatment; MIP | Treatment as Usual at Child Health Centres
Number analyzed (Participants) | 38 | 37
Scores on a scale | 0.64 (0.12) | 0.57 (0.17)
Statistical Analysis 1: Comparison: Mother-infant Psychoanalytic Treatment; MIP vs Treatment as Usual at Child Health Centres; see under the PIR-GAS; Test type: Superiority or Other; p = .031, Regression, Linear; Degrees of freedom (df) = 61.2; Mean Difference (Net) = -0.84, 95% CI 2-sided [-1.61 to -0.08], Standard Error of Mean 0.38

6. Secondary Outcome: General Severity Index of the Symptom Check List-90
Description: The Symptom Check List-90 (SCL-90; Derogatis, 1994), with a Swedish language version (Fridell, Cesarec, Johansson, & Malling Thorsen, 2002), is a self-report questionnaire containing 90 items rated from 0 to 4. Higher scores indicate a worse outcome. The General Severity Index (GSI, or the mean across all items) was used to measure maternal general psychological distress.
Time Frame: two assessments at six month-interval
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Mother-Infant Psychoanalytic Treatment;MIP | Treatment as Usual at Child Health Centre
Number analyzed (Participants) | 38 | 37
Scores on a scale | 0.57 [0.42 to 0.71] | 0.68 [0.54 to 0.83]
Statistical Analysis 1: Comparison: Mother-Infant Psychoanalytic Treatment;MIP vs Treatment as Usual at Child Health Centre; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .158, Mixed Models Analysis; Degrees of freedom (df) = 71.2; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.05 to 0.31], Standard Error of Mean 0.09

ADVERSE EVENTS:
Time Frame: 6 months
Description: Mothers were invited to contact the investigator about any adverse events. The follow-up interviews 6 months after the first thoroughly investigated adverse effects.
Arm/Group | Mother-Infant Psychoanalytic Treatment;MIP | TAU at Child Health Centres
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 0/38 | 0/37

LIMITATIONS AND CAVEATS:
The assumption that assignment to Treatment As Usual (TAU) at Child Health Centres (CHC) would generate disappointment was contradicted: pre-treatment data were more optimal in this group. The final number of non-completers was roughly equal in the two treatment groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No